CLINICAL TRIAL: NCT02105467
Title: A Phase III Randomized Clinical Trial to Study the Efficacy and Safety of the Combination Regimen of MK-5172/MK-8742 in Treatment-Naïve Subjects With Chronic HCV GT1, GT4, and GT6 Infection.
Brief Title: Study of Efficacy and Safety of Grazoprevir (MK-5172)/Elbasvir (MK-8742) Combination Regimen for Treatment-Naïve Participants With Chronic Hepatitis C Virus Genotypes 1, 4, and 6 (MK-5172-060)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5172-060; 2014-000137-22 (EudraCT Number)
Record Dates: First submitted 2014-04-02; First posted 2014-04-07 (Estimated); Results first posted 2016-04-12 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Chronic Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — grazoprevir; elbasvir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Treatment Group (Experimental): Participants received blinded grazoprevir 100 mg / elbasvir 50 mg fixed-dose combination (FDC) tablet orally once daily for 12 weeks followed by a 24-week follow-up period
  Interventions: Drug: Grazoprevir 100mg / Elbasvir 50 mg FDC
- Deferred Treatment Group (Placebo Comparator): Participants received blinded placebo tablet orally once daily for 12 weeks; after a 4-week unblinding/washout period participants received open label grazoprevir 100 mg / elbasvir 50 mg FDC tablet orally once daily for 12 weeks. Follow-up was continued for an additional 24 weeks.
  Interventions: Drug: Grazoprevir 100mg / Elbasvir 50 mg FDC; Drug: Placebo to Grazoprevir / Elbasvir 50 mg FDC

INTERVENTIONS:
Drug: Grazoprevir 100mg / Elbasvir 50 mg FDC
Drug: Placebo to Grazoprevir / Elbasvir 50 mg FDC
  Arms: Deferred Treatment Group

SUMMARY:
This was an efficacy and safety study of grazoprevir (MK-5172) in combination with elbasvir (MK-8742) in treatment-naive participants with chronic hepatitis C virus (HCV) genotype (GT) 1, 4, or 6 infection. Participants were randomly assigned (3:1 ratio) to immediate treatment or deferred treatment (placebo control). The primary efficacy hypothesis was that the proportion of participants receiving combination therapy in the Immediate Treatment Arm who achieve sustained viral response at 12 weeks after the end of study treatment (SVR12) is superior to 73%.

ELIGIBILITY:
Inclusion criteria:

* Documented chronic HCV GT1, GT4, or GT6 with no evidence of non-typeable or mixed genotype infection (positive for anti-HCV antibody, HCV RNA, or any of the listed GTs at least 6 months prior to screening must be confirmed by screening lab results)
* Cirrhosis defined by: liver biopsy showing cirrhosis METAVIR F4; or Fibroscan showing cirrhosis with a result of >12.5 kiloPascals (kPa); or FibroSure® (Fibrotest®) score of >0.75 and an aspartate aminotransferase (AST): platelet ratio index (APRI) of >2
* Absence of cirrhosis defined by: liver biopsy showing absence of cirrhosis, or Fibroscan with a result of ≤12.5 kPa, or Fibrosure® (Fibrotest®) score of <= 0.48 and APRI of <=1
* HCV treatment status of treatment naïve (naïve to all anti-HCV treatment) and can also be ineligible to take pegylated interferon
* Female participant not of reproductive potential, or female of reproductive potential and agrees to avoid becoming pregnant while receiving study drug and for 14 days after the last dose of study drug (using abstinence or acceptable methods of contraception)

Exclusion criteria:

* Evidence of decompensated liver disease manifested by the presence of or history of ascites, esophageal or gastric variceal bleeding, hepatic encephalopathy or other signs or symptoms of advanced liver disease. For cirrhotics, participants who are Child-Pugh Class B or C or who have a Pugh-Turcotte (CPT) score >6
* Co-infection with hepatitis B virus or human immunodeficiency virus (HIV)
* History of malignancy <=5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer or carcinoma in situ; or is under evaluation for other active or suspected malignancy
* Evidence of hepatocellular carcinoma (HCC) or under evaluation for HCC
* Currently participating or has participated in a study with an investigational compound within 30 days of signing informed consent and is not willing to refrain from participating in another such study during the course of this study
* Clinically-relevant drug or alcohol abuse within 12 months of screening
* Pregnant, breast-feeding, or expecting to conceive or donate eggs from Day 1 throughout treatment and 14 days after the last dose of study medication or longer if dictated by local regulations
* Organ transplant (including hematopoietic stem cell transplants) other than cornea and hair
* Poor venous access
* History of gastric surgery (e.g., stapling, bypass) or history of malabsorption disorder (e.g., celiac sprue disease)
* Any medical condition requiring, or likely to require, chronic systemic administration of corticosteroids, TNF antagonists, or other immunosuppressant drugs during the course of the trial
* Evidence of history of chronic hepatitis not caused by HCV, including but not limited to nonalcoholic steatohepatitis (NASH), drug-induced hepatitis, and autoimmune hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2014-06-05 (Actual); Primary Completion 2015-02-26 (Actual); Study Completion 2015-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Zeuzem S, Ghalib R, Reddy KR, Pockros PJ, Ben Ari Z, Zhao Y, Brown DD, Wan S, DiNubile MJ, Nguyen BY, Robertson MN, Wahl J, Barr E, Butterton JR. Grazoprevir-Elbasvir Combination Therapy for Treatment-Naive Cirrhotic and Noncirrhotic Patients With Chronic Hepatitis C Virus Genotype 1, 4, or 6 Infection: A Randomized Trial. Ann Intern Med. 2015 Jul 7;163(1):1-13. doi: 10.7326/M15-0785. PMID 25909356
- [Derived] Asselah T, Reesink H, Gerstoft J, de Ledinghen V, Pockros PJ, Robertson M, Hwang P, Asante-Appiah E, Wahl J, Nguyen BY, Barr E, Talwani R, Serfaty L. Efficacy of elbasvir and grazoprevir in participants with hepatitis C virus genotype 4 infection: A pooled analysis. Liver Int. 2018 Sep;38(9):1583-1591. doi: 10.1111/liv.13727. Epub 2018 Mar 31. PMID 29461687
- [Derived] Reau N, Robertson MN, Feng HP, Caro L, Yeh WW, Nguyen BT, Wahl J, Barr E, Hwang P, Klopfer SO. Concomitant proton pump inhibitor use does not reduce the efficacy of elbasvir/grazoprevir: A pooled analysis of 1,322 patients with hepatitis C infection. Hepatol Commun. 2017 Aug 22;1(8):757-764. doi: 10.1002/hep4.1081. eCollection 2017 Oct. PMID 29404492
- [Derived] Jacobson IM, Lawitz E, Kwo PY, Hezode C, Peng CY, Howe AYM, Hwang P, Wahl J, Robertson M, Barr E, Haber BA. Safety and Efficacy of Elbasvir/Grazoprevir in Patients With Hepatitis C Virus Infection and Compensated Cirrhosis: An Integrated Analysis. Gastroenterology. 2017 May;152(6):1372-1382.e2. doi: 10.1053/j.gastro.2017.01.050. Epub 2017 Feb 11. PMID 28193518

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For Subject Disposition, Period 1 covers Day 1 through Week 12 for both treatment groups. Period 2 covers Week 12 through Week 36 for the Immediate Treatment Group (ITG) and Week 12 through Week 28 for the Deferred Treatment Group (DTG). Period 3 covers Week 28 through Week 52 for the DTG; the ITG completed the study with Period 2.
Pre-assignment Details: A total of 469 participants were screened and 421 were randomized.
Groups:
- Immediate Treatment Group: Participants received blinded grazoprevir 100 mg / elbasvir 50 mg fixed-dose combination (FDC) tablet orally once daily for 12 weeks (Period 1), followed by a 24-week follow-up period (Period 2)
- Deferred Treatment Group: Participants received blinded placebo tablet orally once daily for 12 weeks (Period 1), followed by a 4-week unblinding/washout period and 12 weeks of open label grazoprevir 100 mg / elbasvir 50 mg FDC tablet orally once daily (Period 2), followed by a 24-week follow-up period (Period 3).
Period: Period 1
Arm/Group | Immediate Treatment Group | Deferred Treatment Group
Started | 316 | 105
Completed | 314 | 105
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 1 | 0
Period: Period 2
Arm/Group | Immediate Treatment Group | Deferred Treatment Group
Started | 314 | 104 (One participant did not receive deferred treatment (Period 2) but proceeded directly to Period 3)
Completed | 312 | 102
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Period: Period 3
Arm/Group | Immediate Treatment Group | Deferred Treatment Group
Started | 0 (The Immediate Treatment Group completed the study with Period 2) | 103 (One participant did not receive deferred treatment (Period 2) but proceeded directly to Period 3)
Completed | 0 | 102
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Deferred Treatment Group: Participants received blinded placebo tablet orally once daily for 12 weeks; after a 4-week unblinding/washout period participants received open label grazoprevir 100 mg / elbasvir 50 mg FDC tablet orally once daily for 12 weeks. Follow-up was for an additional 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Immediate Treatment Group | Deferred Treatment Group | Total
Number analyzed (Participants) | 316 | 105 | 421
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.2 (11.1) | 53.8 (11.2) | 52.6 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 49 | 194
  Male | 171 | 56 | 227
HCV Genotype [Number; unit: Participants]
  Genotype 1a | 157 | 54 | 211
  Genotype 1b | 131 | 40 | 171
  Genotype 4 | 18 | 8 | 26
  Genotype 6 | 10 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virologic Response at 12 Weeks After the End of Treatment (SVR12)
Description: Hepatitis C Virus (HCV) ribonucleic acid (RNA) was measured using the Roche COBAS® Taqman® HCV Test, v2.0 assay. SVR12 was defined as HCV RNA <Lower Limit of Quantification (<15 IU/mL) 12 weeks after the end of all study therapy.
Time Frame: Week 24 (12 weeks after the end of treatment)
Population: The Full Analysis Set included randomized participants who received at least one dose of study treatment. This outcome measure applied only to the Immediate Treatment group.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Immediate Treatment Group
Number analyzed (Participants) | 316
Percentage of participants | 94.6 [91.5 to 96.8]
Statistical Analysis 1: Comparison: Immediate Treatment Group; Superiority of SVR12 in the Immediate Treatment group was tested against the historical response rate of 73%; Test type: Superiority or Other; p < 0.001, One-sided, one-sample exact test

2. Primary Outcome: Percentage of Participants Experiencing at Least One Adverse Event
Description: An adverse event is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an adverse event.
Time Frame: Up to Week 14 (14 days after the Blinded Treatment was completed)
Population: The All Subjects as Treated population included randomized participants who received at least one dose of study treatment. This outcome measure applied only to the blinded treatment period.
Measure: Number; unit: Percentage of participants
Arm/Group | Immediate Treatment Group | Deferred Treatment Group
Number analyzed (Participants) | 316 | 105
Percentage of participants | 67.4 | 68.6
Statistical Analysis 1: Comparison: Immediate Treatment Group vs Deferred Treatment Group; Test type: Superiority or Other; Risk Difference (RD) = -1.0, 95% CI 2-sided [-10.8 to 9.6] — Between-treatment difference (Immediate Treatment Group - Deferred Treatment Group) was analyzed using the Miettinen and Nurminen method

3. Primary Outcome: Percentage of Participants Discontinued From Study Treatment Because of an Adverse Event
Description: as for outcome 2
Time Frame: Up to Week 12 (end of Blinded Treatment)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Immediate Treatment Group | Deferred Treatment Group
Number analyzed (Participants) | 316 | 105
Percentage of participants | 0.9 | 1.0
Statistical Analysis 1: Comparison: Immediate Treatment Group vs Deferred Treatment Group; Test type: Superiority or Other; Risk Difference (RD) = -0.0, 95% CI 2-sided [-4.4 to 2.0] — [estimate comment as in outcome 2, analysis 1]

4. Other Pre Specified Outcome: Percentage of Participants Achieving Sustained Virologic Response at 4 Weeks After the End of Treatment (SVR4)
Description: Hepatitis C Virus RNA was measured using the Roche COBAS® Taqman® HCV Test, v2.0 assay. SVR4 was defined as HCV RNA <Lower Limit of Quantitation (<15 IU/mL) 4 weeks after the end of all study therapy.
Time Frame: Week 16 (4 weeks after the end of treatment)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Immediate Treatment Group
Number analyzed (Participants) | 316
Percentage of participants | 97.2 [94.7 to 98.7]

5. Secondary Outcome: Percentage of Participants Achieving Sustained Virologic Response at 24 Weeks After the End of Treatment (SVR24)
Description: Hepatitis C Virus RNA was measured using the Roche COBAS® Taqman® HCV Test, v2.0 assay. SVR24 was defined as HCV RNA <Lower Limit of Quantitation (<15 IU/mL) 24 weeks after the end of all study therapy.
Time Frame: Week 36 (24 weeks after the end of treatment)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Immediate Treatment Group
Number analyzed (Participants) | 316
Percentage of participants | 94.3 [91.1 to 96.6]

ADVERSE EVENTS:
Time Frame: Immediate Treatment Group: Up to Week 36; Deferred Treatment Group (Blinded Treatment): Up to Week 16; Deferred Treatment Group (Open-label Treatment): Week 16 to Week 52
Groups:
- Immediate Treatment Group: Participants received blinded grazoprevir 100 mg / elbasvir 50 mg fixed-dose combination (FDC) tablet orally once daily for 12 weeks followed by a 24-week follow-up period. Adverse event reporting covers Day 1 through Week 36.
- Deferred Treatment Group (Blinded Treatment): Participants received blinded placebo tablet orally once daily for 12 weeks; after a 4-week unblinding/washout period participants received open label grazoprevir 100 mg / elbasvir 50 mg FDC tablet orally once daily for 12 weeks. Follow-up was for an additional 24 weeks. Adverse event reporting covers Day 1 through Week 16.
- Deferred Treatment Group (Open-label Treatment): Participants received blinded placebo tablet orally once daily for 12 weeks; after a 4-week unblinding/washout period participants received open label grazoprevir 100 mg / elbasvir 50 mg FDC tablet orally once daily for 12 weeks. Follow-up was for an additional 24 weeks. Adverse event reporting covers Week 16 through Week 52.
Arm/Group | Immediate Treatment Group | Deferred Treatment Group (Blinded Treatment) | Deferred Treatment Group (Open-label Treatment)
Serious Adverse Events (participants affected / at risk) | 15/316 | 4/105 | 3/103
Other Adverse Events (participants affected / at risk) | 147/316 | 60/105 | 42/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Treatment Group (N=316) | Deferred Treatment Group (Blinded Treatment) (N=105) | Deferred Treatment Group (Open-label Treatment) (N=103)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hiatus hernia strangulated (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Peritoneal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Treatment Group (N=316) | Deferred Treatment Group (Blinded Treatment) (N=105) | Deferred Treatment Group (Open-label Treatment) (N=103)
Diarrhoea (Gastrointestinal disorders) | 14 (15) | 7 (7) | 5 (5)
Nausea (Gastrointestinal disorders) | 29 (32) | 8 (8) | 8 (8)
Fatigue (General disorders) | 49 (53) | 18 (19) | 12 (13)
Nasopharyngitis (Infections and infestations) | 20 (23) | 7 (8) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (22) | 6 (6) | 3 (3)
Dizziness (Nervous system disorders) | 9 (9) | 7 (9) | 0 (0)
Headache (Nervous system disorders) | 51 (61) | 18 (19) | 17 (19)
Insomnia (Psychiatric disorders) | 6 (6) | 6 (6) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (7) | 8 (9) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 17 (18) | 2 (2) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 3 (3) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.